CLINICAL TRIAL: NCT07113496
Title: An Exploratory Clinical Study on the Safety and Efficacy of Allogeneic CAR-T Cell (RN1201) for Relapsed/Refractory CD19+/BCMA+ Hematologic Malignancies
Brief Title: RN1201injection for Relapsed/Refractory CD19+/BCMA+ Hematologic Malignancies
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Lei Fan, Director of lymphoma center, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN1201-Onc
Record Dates: First submitted 2025-07-24; First posted 2025-08-08 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Relapsed or Refractory B-cell Hematologic Malignancies; B-cell Acute Lymphoblastic Leukemia (B-ALL); Multiple Myeloma (MM); Plasmablastic Lymphoma; Relapsed or Refractory CD19+/BCMA+ Hematologic Malignancies; Mature B-Cell Lymphoma
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma; Multiple Myeloma; Plasmablastic Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic CAR-T cell therapy (Experimental): RN1201 cells injection will be infused via intravenously
  Interventions: Biological: Allogeneic CAR-T

INTERVENTIONS:
Biological: Allogeneic CAR-T — Patients will receive lymphodepletion chemotherapy followed by a single intravenous infusion of Allogeneic CAR-T cells. In select cases, CAR-T infusion may be administered post-autologous hematopoietic stem cell transplantation (auto-HSCT)

SUMMARY:
This single-arm, dose-escalation exploratory trial evaluates the safety and efficacy of Allogeneic CAR-T (UCAR-T) cell therapy in patients with relapsed or refractory CD19+/BCMA+ hematologic malignancies, including those with minimal residual disease (MRD). Eligible patients will receive lymphodepletion followed by a single infusion of UCAR-T cells, either post-transplant or without transplantation depending on disease status. The trial assesses overall response and disease control rates, treatment-emergent adverse events, and in vivo behavior of UCAR-T cells.

DETAILED DESCRIPTION:
This single-arm, dose-escalation exploratory trial evaluates the safety and efficacy of Allogeneic CAR-T (UCAR-T) cell therapy in patients with relapsed or refractory CD19+/BCMA+ hematologic malignancies, including those with minimal residual disease (MRD). Eligible patients will receive lymphodepletion followed by a single infusion of UCAR-T cells, either post-transplant or without transplantation depending on disease status.Primary endpoints include treatment-emergent adverse events (TEAEs) and dose-limiting toxicities (DLTs). Secondary endpoints include objective response rate (ORR), disease control rate (DCR), pharmacokinetics, and pharmacodynamics of UCAR-T. This study aims to provide initial evidence for the safety and anti-tumor activity of UCAR-T in CD19+/BCMA+ hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria

1. Voluntary participation with signed informed consent.
2. Pathologically confirmed CD19-positive and/or B-cell maturation antigen (BCMA)-positive hematologic malignancy according to the WHO 2017 classification, including but not limited to multiple myeloma, B-cell acute lymphoblastic leukemia (B-ALL), mature B-cell lymphomas, and plasmablastic lymphoma.
3. Relapsed/refractory disease defined as failure to achieve complete remission after standard therapy, or relapse after an initial response during treatment or follow-up.
4. Measurable disease required:

   1. For B-ALL: persistent minimal residual disease (MRD) positivity despite hematologic remission.
   2. For lymphoma: at least one measurable lesion ≥1.5 cm in longest diameter per IWG revised criteria.
   3. For multiple myeloma: positive immunofixation electrophoresis or presence of extramedullary disease.
5. Age ≥18 years; both sexes eligible.
6. Expected survival ≥12 weeks.
7. Adequate organ function (exceptions for disease-related impairment are at the investigator's discretion):

   1. Total bilirubin <2× upper limit of normal (ULN); serum creatinine <ULN; ALT and AST <3× ULN.
   2. Absolute neutrophil count ≥0.5×10⁹/L; platelets ≥20×10⁹/L (no requirement if marrow involvement is documented).
   3. Eastern Cooperative Oncology Group (ECOG) performance status 0-3.
   4. Left ventricular ejection fraction (LVEF) ≥50%.

Exclusion Criteria

1. Known hypersensitivity, allergy, intolerance, or contraindication to CD19/BCMA-UCAR-T or any study drugs (fludarabine, cyclophosphamide, tocilizumab).
2. Genetic syndromes: Fanconi, Kostmann, Shwachman, or any documented bone-marrow failure syndrome.
3. Active or uncontrolled infection requiring IV antibiotics; evidence of severe active infection.
4. NYHA Class III or IV heart failure (unless clearly secondary to the underlying malignancy).
5. Central Nervous System (CNS) disorders unrelated to the primary hematologic malignancy.
6. Prior malignancy except adequately treated carcinoma in situ of skin, cervix, lung, or other non-active tumors.
7. Significant bleeding diathesis (e.g., gastrointestinal (GI) bleeding, coagulopathy, hypersplenism).
8. History of significant cardiac disease within the past 3 months that, in the investigator's judgment, renders the patient unable to tolerate study participation..
9. Pregnancy, lactation, or planned pregnancy within 6 months.
10. Any condition that, in the investigator's opinion, may increase risk or interfere with study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events (TEAEs) and dose-limiting toxicities (DLTs) | DLTs: Within 28 days after CAR-T cell infusion; TEAEs: From infusion up to 12 months post-treatment.
  TEAEs and DLTs will be graded according to CTCAE v5.0 and ASTCT consensus criteria

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Week 4, Month 3, Month 6 and Month 12
  Identify the number of patients with complete response (CR), Identify the number of patients with partial response (PR), and Calculate ORR=(CR+PR)/total patients
Disease control rate (DCR) | Week 4, Month 3, Month 6 and Month 12
  Identify the number of patients with complete response (CR), partial response (PR), stable disease (SD) and calculate DCR=(CR+PR+SD)/total patients
Progression-free survival (PFS) | Week 4, Month 3, Month 6 and Month 12
  PFS defned as the time from the date of RN1201 infusion to the frst assessment of confrmed disease progression or death
Overall survival (OS) | Week 4, Month 3, Month 6 and Month 12
  OS defned as the time from the date of RN1201 infusion to death
Cmax of RN1201 | Up to 12 months
  peak plasma concentration of CAR - T cells copy number and the positive rate
Tmax of RN1201 | Up to 12 months
  Time to maximum concentration of RN1201
Cytokines in the peripheral blood after RN1201 infusion | Up to 12 months
  Serum concentrations of interleukin (IL)-2, IL-6, IL-8, IL-10, interferon-gamma (IFN-γ), and TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Lei Fan, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No